CLINICAL TRIAL: NCT05747105
Title: A 16-Week Sleep Extension Pilot Study in Adults With Obesity
Brief Title: A Sleep Extension Pilot Study in Adults With Obesity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to move forward with the study due to personnel changes
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 852866
Record Dates: First submitted 2023-02-06; First posted 2023-02-28 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Sleep; Weight, Body; Eating Behavior; Blood Pressure; Quality of Life
Keywords: short sleep duration; sleep extension; obesity; eating behavior; blood pressure
MeSH Terms: conditions — Obesity; Body Weight; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This study is a single-arm pilot intervention study to assess the efficacy of a 16-week sleep extension protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Extension Intervention (Experimental): All participants will receive the 16-week sleep extension intervention aimed to lengthen nighttime sleep duration by at least 30-60 minutes per night. No prescription for daily calorie/dietary intake or physical activity will be provided in this study, except behaviors consistent with sleep hygiene recommendations.
  Interventions: Behavioral: Sleep Extension

INTERVENTIONS:
Behavioral: Sleep Extension — The 16-week protocol includes 11 total individual visits that integrate applicable elements of Cognitive Behavioral Therapy for Insomnia (CBT-I) and health behavior change theory. The first 6 weeks include weekly sessions (~45 minutes each) focused on psychoeducation about sleep, goal-setting and self-monitoring, stimulus control, addressing cognitive and somatic arousal, sleep hygiene, and challenging negative thoughts about sleep. Sleep restriction will also be used in specific cases where sleep efficiency is low (<85%). The remaining 10 weeks include briefer biweekly visits (5 visits, ~15-20 minutes each) to reinforce health behavior change strategies through topics such as problem-solving barriers, utilizing social support, identifying setbacks and creating an action plan, and relapse prevention. Self-reported sleep diary data and subjective sleepiness will be collected at each visit.

SUMMARY:
The pilot study will test the feasibility of a 16-week sleep extension intervention, in adults with obesity, to increase nighttime sleep duration, as well as reduce daytime sleepiness and sleep-related disturbance. The study will also examine changes in weight, eating behaviors, wellbeing, and blood pressure across the 16-week intervention .

DETAILED DESCRIPTION:
Short sleep duration (<6.5 hours per night) is a risk factor for poorer health outcomes,1 including overweight and obesity,2 likely due, in part, to its impact on energy intake and eating behaviors. Previous research with experimental sleep restriction and observational studies of short sleepers has shown that short sleep duration is associated with higher calorie intake (including greater calories from fat), increased hunger ratings, a greater number of daily eating occasions, and consumption of larger food portion sizes.3 Short sleep duration is also related to cardiovascular risk factors, including hypertension.4 Sleep extension studies provide some evidence that increasing time spent asleep at night may improve weight, eating behaviors (e.g., net reduction of 270 kcal/d and 0.87 kg over 4 weeks5), and cardiovascular outcomes (e.g., blood pressure6); however, the current literature is limited by short-term intervention and study periods (e.g., 2 to 9 weeks). Therefore, it is unclear if the effects of sleep extension can be sustained over time and if a longer intervention can produce clinically meaningful weight reduction and associated health improvements in adults with obesity. This pilot study will determine the feasibility of a longer, 16-week sleep extension intervention to increase nighttime sleep duration among 10 adults, aged 18-50 years old, with obesity (BMI > 30 kg/m2). Additional secondary outcomes of changes in weight, eating behaviors, wellbeing, and blood pressure will also be assessed. If results are positive, the protocol will be used to secure external funding for a larger randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18-50 years old,
2. All genders
3. Body Mass Index within the obese weight status (BMI of ≥ 30 kg/m2)
4. Short sleep duration, defined as sleeping, on average, <6.5 hours/night for at least 5 nights/week
5. Sleep patterns must be stable for the past 6 months
6. Weight must be stable (+/- 10 lb) for the past 6 months
7. If taking medication for medical or mental health conditions, the condition must be well-controlled with stable dosage (i.e., at least 3 months)
8. Note: Individuals with and without insomnia will be eligible to participate to increase generalizability of the findings. Also, individuals with known obstructive sleep apnea that is being treated and individuals who fall below the "very high risk" category for obstructive sleep apnea (on the ARES screening questionnaire) will be included.
9. Participants must provide a completed form for study participation from their primary care provider to confirm that it is safe from a medical perspective

Exclusion Criteria:

1. Specific chronic sleep disorders (e.g., untreated or at very high risk for obstructive sleep apnea, restless leg syndrome, parasomnias, narcolepsy, central apnea, chronic fatigue syndrome, or fibromyalgia)
2. Extreme chronotype (i.e., extreme morning or evening sleep patterns)
3. Work schedule that is not compatible with sleep habit changes (e.g., night shifts, rotating shift work, or long driving)
4. Chronic use of sleep aid or anticonvulsant medications
5. Chronic organ disorders (e.g., untreated or uncontrolled diabetes, other endocrine disorders, COPD, chronic cardiac arrhythmia, uncontrolled hypertension or gastro-esophageal disorders)
6. Current enrollment in a weight loss program or any active weight loss attempt (e.g., self-directed diet/exercise, over-the-counter supplements, weight management medication)
7. History of bariatric surgery (with the exception of an adjustable gastric band that has been removed)
8. Mental health disorders judged severe (e.g., major depression, eating disorders, anxiety disorders, bipolar disorder/mania, schizophrenia, active suicidal ideation)
9. Substance use (e.g., illicit drugs, marijuana dependence, excessive caffeine intake, smoking/tobacco use)
10. Planned move outside of the Philadelphia area in the next 6 months
11. Planned travel across time zones during the study period
12. Family factors that may interfere with adherence to the study protocol (e.g., infants and young children that consistently disrupt their sleep schedule; partner, other individuals, or pets that would make compliance difficult)
13. Pregnancy or lactation or plans to become pregnant during the study period
14. Menopause
15. Any other contraindication to participation as determined by the study team

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of intervention session attendance | Baseline to Week 16 of the intervention
  The percentage of sessions attended by participants across the 16-week intervention
Percentage of participants who complete the study | Baseline to Week 16 of the intervention
  The percentage of participants who complete the final Week 16 visit

SECONDARY OUTCOMES:
Change in nighttime sleep duration | Baseline to Week 16 of the intervention
  Average nighttime sleep duration as measured by actigraphy during a 1-week monitoring period
Change in weight | Baseline to Week 16 of the intervention
  Weight as measured in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, Ph.D., Principal Investigator — University of Pennsylvania; Philip Gehrman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No